CLINICAL TRIAL: NCT06575322
Title: Effects of Neoadjuvant Therapy With Carboplatin, Paclitaxel Combined With Anti-PD-1 Drugs on Pain, Anxiety and Depression in Patients With Resectable Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Song Fan, MD, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-646-01
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant therapy+ Surgery group( Group A): The patient was diagnosed with head and neck squamous cell carcinoma (stage I-IVA), untreated, and planned to undergo surgical treatment + combined chemotherapy and immunotherapy.
  Interventions: Drug: Carboplatin（ neoadjuvant）; Drug: Paclitaxel （neoadjuvant）; Drug: Anti-PD-1 Drugs; Procedure: Surgical resection
- Direct surgery group (Group B): The patient was diagnosed with head and neck squamous cell carcinoma (stage I-IVA), untreated, and planned to undergo surgery.
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Drug: Carboplatin（ neoadjuvant） — Carboplatin (IV), AUC=5，administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Groups: Neoadjuvant therapy+ Surgery group( Group A)
Drug: Paclitaxel （neoadjuvant） — Nab-paclitaxel 260mg/m2 administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Groups: Neoadjuvant therapy+ Surgery group( Group A)
Drug: Anti-PD-1 Drugs — Anti-PD-1 Drugs 200 mg administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Groups: Neoadjuvant therapy+ Surgery group( Group A)
Procedure: Surgical resection — Standard of care

SUMMARY:
The goal of this observational study is to learn about the Effects of neoadjuvant therapy with carboplatin, paclitaxel combined with anti-PD-1 drugs on pain, anxiety and depression in patients with operable head and neck squamous cell carcinoma: a prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

- 1: Clinical diagnosis of head and neck squamous cell carcinoma (stage I-IVA), without prior treatment, and planning to undergo either surgical treatment alone or surgical treatment combined with chemotherapy and immunotherapy.

2: Ability to speak Chinese and possess basic reading and writing skills.

Exclusion Criteria:

* 1: Presence of mental illnesses such as dementia or delirium.

  2: Active use of narcotic drugs, including consuming alcohol more than 4 times per day or more than 4 times per week.

  3: Patients who alter their treatment plan during the course of treatment.

  4: Current or prior use of antidepressants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were diagnosed with head and neck squamous cell carcinoma (stages I-IV) and did not receive treatment. They planned to receive only surgical treatment or combined surgical treatment + chemotherapy and immunotherapy. They were divided into two groups, and the participating groups were selected according to the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (Short Form) | Baseline, 9 weeks, 6 months, 12 months
  The BPI-SF contains 15 items that measure pain severity and pain interference, with each item assessed on an 11-point numeric rating scale ranging from "no pain" (0) to "worst pain imaginable" (10).
HADS | Baseline, 9 weeks, 6 months, 12 months
  HADS is a 14-item self-report scale, including two subscales: anxiety (HADS-A) and depression (HADS-D). The total HADS score ranges from 0 to 42, and the subscales range from 0 to 21.

SECONDARY OUTCOMES:
Major pathological response rate | Within 30 days after surgery
  Defined as the proportion of subjects with ≤10% viable tumor cells in resection specimens to total subjects
Complete pathological response rate | Within 30 days after surgery
  Defined as the proportion of subjects without viable tumor cells in the resection specimen to the total subjects

CONTACTS AND LOCATIONS:
Overall Officials: Song Fan, Doctor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guanzhou, Guangdong, China